CLINICAL TRIAL: NCT02180919
Title: Implementation of Telemonitoring in the Management of Acute Exacerbations of Chronic Heart Failure and Respiratory Failure/Chronic Obstructive Pulmonary Disease
Brief Title: Implementation of Telemonitoring in Chronic Heart or Lung Failure
Acronym: TELECRAFT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 10/H0704/19; 10/H0704/19 (Other: Royal Brompton Hospital REC/research office)
Record Dates: First submitted 2014-06-19; First posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2010-05

CONDITIONS: COPD; Heart Failure; Respiratory Failure
Keywords: Telemonitoring; COPD; Heart failure; Exacerbation; Respiratory failure; Prevention; Self monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control period (No Intervention): All patients with receive standard optimal medical care according to ESC Heart Failure guidelines, NICE COPD guidelines or other best practice care pathways as relevant to their condition.
- Telemonitoring (Experimental): telemonitoring will be carried out in the patient's home using the conformity European (CE) marked Philips Motiva system which comprises weight scales, blood pressure and heart rate monitoring, finger pulse oximeter and provides question/answer prompts all of which is linked to the patient's television screen and can be tuned into just as like a television (TV) channel. Measurements of blood pressure, heart rate and weight will be obtained from the heart failure patients daily. In the respiratory patients heart rate and oximetry will be measured daily, and blood pressure and weight once a week.
  Interventions: Device: CE marked Philips Motiva system

INTERVENTIONS:
Device: CE marked Philips Motiva system — Telemonitoring will be carried out in the patient's home using the CE marked Philips Motiva system which comprises weight scales, blood pressure and heart rate monitoring, finger pulse oximeter and provides question/answer prompts all of which is linked to the patient's television screen and can be tuned into just as like a TV channel. Measurements of blood pressure, heart rate and weight will be obtained from the heart failure patients daily. In the respiratory patients heart rate and oximetry will be measured daily, and blood pressure and weight once a week.
  Arms: Telemonitoring

SUMMARY:
The aims of the study are to:

1. Implement a telemonitoring programme in heart failure and obstructive pulmonary disease (COPD) /chronic respiratory patients by assessing the real world impact of on readmissions, consults, home visits, quality of life and economic endpoints.
2. Explore the effects of telemonitoring across heart and respiratory groups with respect to i) factors that influence how patients integrate telemonitoring into their daily routines and self care behaviour and ii) how healthcare professionals use telemonitoring to aid decision- making.
3. Understand the impact of telemonitoring on a variety of care pathways.

DETAILED DESCRIPTION:
BACKGROUND

Heart failure exacerbations consume 60-70% of costs for the condition and COPD exacerbations lead to 1:8 admissions so are costly to the NHS. The roll-out of telemonitoring in chronic disease is in line with NHS policy (Building Telecare in England; High Quality Care for All, national health service (NHS) next stage Darzi review).

Despite systematic reviews, the Whole System Demonstrator programme and randomised control trial (RCT) evidence in heart failure, the outcome of implementing telemonitoring is unclear, the evidence base in COPD is less consistent, and few studies have included economic analysis or investigated cross speciality implementation. An Italian trial found that telemedicine reduces chronic respiratory admissions by a third, but the Italian health service differs from the united kingdom (UK) system. The european union (EU) Commission Communication on telemedicine 2009 has stressed the need for new deployments to contribute to the evidence base in respiratory disease, and include a detailed analysis of the process changes that determine success. Our group has previously shown that telemonitoring reduces unplanned admissions in heart failure patients, and that elderly patients were able to cope well with the equipment. The investigators have also had experience with telesupport in chronic respiratory patients.

RATIONALE FOR CURRENT STUDY

The study will assess the implementation of a telemonitoring programme to demonstrate

1. whether home telemonitoring alerts patients and health professionals to exacerbations and reduces admissions,
2. if it can be reasonably implemented cross specialty,
3. the impact on quality of life of patients,
4. interaction between healthcare professionals, robustness of algorithms and self efficacy in patients.

The cross-over design allows sustained effects on self care and admissions to be assessed after removal of telemonitoring at 6 months in first groups treated. The acceptability of telemonitoring to healthcare workers and factors aiding and limiting integration into care pathways will be explored. Results should inform the commissioning of telemonitoring locally/nationally, facilitate buy-in from secondary and primary care teams, and optimise cost.

OVERALL DESIGN

Design: Crossover implementation study with patients allocated randomly 1:1 to telemonitoring or delayed entry to telemonitoring (after 6 months). All patients with receive standard optimal medical care according to European Society of Cardiology (ESC) Heart Failure guidelines, National Institute for Health and Care Excellence (NICE) COPD guidelines or other best practice care pathways as relevant to their condition. Each patient will receive home telemonitoring for 6 months. Comparisons will be carried out between patients with delayed entry (controls) and active telemonitoring. In the group receiving telemonitoring in first 6 month period the investigators will be able to assess impact of withdrawal in subsequent 6 months ie longer term benefit.

TELEMONITORING

Data from the monitors are delivered to the health care team members personal computer (PCs) using a dedicated broad band line which is installed in the patients home and is routed via a secure Philips Server. Each patient receives education in using the device until he or she and/or family/carer are fully confident. Via information displayed on their television screen each day patients are requested to answer interactive questions on level of breathlessness, sleep quality, phlegm production, wheeze. These results from each patient is used to create a warning system such that if all parameters are satisfactory this will appear as a green light; or for example, if a drop in arterial oxygen saturation and increase in wheeze, or increase in weight and increased breathlessness is seen the Motiva system will generate a red light for that patient which needs to be acted upon. It is an interactive system and therefore the healthcare team member can advise the patient through their screen (eg. increase dose of diuretic or oxygen flow rate, start antibiotic and steroids), or provide educational material eg. on inhaler use or exercise, and patients can respond. Patients will also be asked several questions once a week on whether they have consulted their general practitioner (GP), visited an Accident and Emergency Dept or been admitted to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients: age > 18 years who were in New York Heart Association class II-IV at time of discharge diagnosed by ESC guidelines.
* Respiratory patients: age > 18 years with diagnosis of COPD or respiratory insufficiency due to chronic respiratory disorder diagnosed by Consultant Respiratory Physician (eg. bronchiectasis, chest wall disease, neuromuscular disorder) and arterial oxygen saturation value during most recent admission for exacerbation of 90% or below (or partial pressure of oxygen in arterial blood (PaO2) 8.0 kilopascal (kPa) or below) on air, or who fulfill criteria for, and receive long term oxygen therapy.

Exclusion Criteria:

* Age <18 years.
* Cognitive impairment sufficient to interfere with use of telemonitoring system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Time to first event | at 6 months
  Acute admission coded as due to acute exacerbation of heart failure/COPD, respiratory failure or mortality from heart failure/respiratory failure/COPD.

SECONDARY OUTCOMES:
Compliance with telemonitoring | averaged over the expected 6 month period
  Daily input into the Motiva system will be collected Monday to Friday. At the end of the study period the compliance with inputting the data on a daily basis will be averaged. This information will provide compliance with telemonitoring data.
Self Efficacy | 0, 3, 6, 9 and 12 months
  The COPD patients will be asked to complete the Bristol COPD Knowledge Questionnaire before and after the 6 month period of telemonitoring, and the heart failure patients invited to complete the Self Care of Heart Failure index before and after telemonitoring.
Focus interviews | 6 and 12 months after completion of the study
  Focus structured interviews will be carried out individually in the patient's home or at Royal Brompton Hospital after 6 and 12 months.
Health care contacts | 0,1,2,3,4,5,6,7,8,9,10,11 and 12 months
  GP consultations, emergency room visits will be recorded monthly in a self reported questionnaire
Hospital Anxiety and Depression Score (HADS) | 0, 3, 6, 9 and 12 months
  The HADS score determines the levels of anxiety and depression that a patient is experiencing. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression.
Minnesota Living with Heart Failure questionnaire | 0, 3, 6, 9 and 12 months
  Minnesota Living with Heart Failure questionnaire measures the effects of symptoms, functional limitations, psychological distress on an individual's quality of life, the Minnesota Living with Heart Failure questionnaire asks each person to indicate using a 6-point, zero to five, Likert scale how much each of 21 facets prevented them from living as they desired
The EuroQOL five dimensions questionnaire (EQ 5D) | 0, 3, 6, 9 and 12 months
  The self-assessment questionnaire is self-reported description of the subject's current health in 5 dimensions i.e., mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The subject is asked to grade their own current level of function in each dimension into one of three degrees of disability (severe, moderate or none).
Chronic Respiratory Disease Questionnaire (CRQ) | 0, 3, 6, 9 and 12 months
  The CRQ is a self-reported, disease specific measurement tool to assess health related quality of life (HRQL) in patients with chronic respiratory disease. Consists of 20 items across four dimensions: dyspnea, fatigue, emotional function, and mastery.

CONTACTS AND LOCATIONS:
Overall Officials: Anita K Simonds, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Brompton Hospital, London
  - West Middlesex University Hospita, London

REFERENCES:
- [Derived] Chatwin M, Hawkins G, Panicchia L, Woods A, Hanak A, Lucas R, Baker E, Ramhamdany E, Mann B, Riley J, Cowie MR, Simonds AK. Randomised crossover trial of telemonitoring in chronic respiratory patients (TeleCRAFT trial). Thorax. 2016 Apr;71(4):305-11. doi: 10.1136/thoraxjnl-2015-207045. PMID 26962013